CLINICAL TRIAL: NCT01931410
Title: The Effect of Rectal and Sublingual Misoprostol Administration in Postpartum or Intrapartum Haemorrhage at Elective Caesarean Delivery: a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, M.D. Obstetric and Gynecology, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Aşıcıoğlu-05
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: ıntrapartum Haemorrhage; Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- sublingual (Placebo Comparator): 400 microgram mısoprostol will be administered sublıngually before elective caesarean
  Interventions: Drug: Misoprostol
- rectal (Placebo Comparator): rectal 600 mgr misoprostol will be administered
  Interventions: Drug: Misoprostol
- synpitan (No Intervention)

INTERVENTIONS:
Drug: Misoprostol
  Arms: rectal; sublingual

SUMMARY:
The investigators hypothesis in this study is that administration of rectal and sublingual misoprostol decreases intrapartum and postpartum haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. live and singleton pregnancy
2. Elective caesarean
3. Gestational week greater than 37 weeks
4. patient between 18-44 year old

Exclusion Criteria:

1. -multiple pregnancy
2. Preeclampsia
3. Gestational diabetes
4. Macrosomia
5. Oligohidraamnıos
6. Polihidraamnıos
7. Myoma
8. Morbid obesity
9. Coagulatıon defect (such as HELLP syndrome)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 618 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Postpartum Haemorrhage | postpartum 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Berhan AŞICIOĞLU, M.D., Principal Investigator — T.C.S.B. Kanuni Sultan Süleyman Research Hospital